CLINICAL TRIAL: NCT07253363
Title: Investigation of Circulating ACTIvin-A and FSTL3 as Prognostic and Predictive BIOmarkers in Precapillary Pulmonary Hypertension
Brief Title: Circulating Activin-A and FSTL3 in Precapillary Pulmonary Hypertension
Acronym: ACTIBIO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP231330; N° IDRCB: 2023-A02244-41 (Registry Identifier: ANSM)
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension; biomarkers; FSTL3; Activin-A
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- No Intervention (Other): No Intervention
  Interventions: Other: Biological collection

INTERVENTIONS:
Other: Biological collection — Serum, plasma, ADN

SUMMARY:
The ACTIOBIO study aims to evaluate the prognostic value of Activin-A and FSTL3 in a large cohort of patients with precapillary pulmonary hypertension, including pulmonary arterial hypertension (Group 1), pulmonary hypertension associated with lung diseases (Group 3), and chronic thromboembolic pulmonary hypertension (Group 4).

DETAILED DESCRIPTION:
In recent years, major advances have been achieved in understanding the cellular and molecular mechanisms underlying pulmonary arterial hypertension (PAH), a major subtype of precapillary PH. These discoveries have led to the development of novel therapeutic strategies, including agents targeting dysregulated pathways of the transforming growth factor beta (TGF-β) superfamily.

Parallel to therapeutic advances, risk stratification at diagnosis and during follow-up has become a cornerstone of PH management. Validated multidimensional tools now integrate clinical, exercise, biomarker, imaging, and hemodynamic parameters to estimate prognosis, guide initial treatment, and define therapeutic goals for follow-up. However, as new therapeutic targets emerge and influence disease trajectory, there is a growing need for novel biomarkers to refine these tools, making them less invasive and more accurate.

Beyond prognostic markers, identifying biomarkers that predict treatment response is essential to move toward precision medicine in PH. Such biomarkers would help tailor therapy to individual patient profiles and optimize long-term outcomes.

The main objective of this study is to analyze the prognostic value of Activin-A and Follistatin-like 3 (FSTL3) in a large cohort of patients with precapillary pulmonary hypertension, including pulmonary arterial hypertension (PAH, group 1), PH associated with lung disease (group 3), and chronic thromboembolic PH (group 4).

ELIGIBILITY:
1. Male or female ≥ 18 years of age
2. Precapillary PH documented by right heart catheterization:

   * mean pulmonary arterial pressure (mPAP) > 20 mmHg,
   * pulmonary artery wedge pressure (PAWP) ≤ 15 mmHg;
   * pulmonary vascular resistance (PVR) > 2 WU
3. Pulmonary arterial hypertension (group 1) or PH associated with lung disease (group 3) or chronic thromboembolic PH (group 4)
4. Patient registered in the French PH registry
5. Patient capable of understanding the study procedures
6. Affiliation to a social security regime (or exemption)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Lung-transplant-free survival at 2 years | Two years
  The primary endpoint is time fto lung-transplantation or death within two years following inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Laurent SAVALE, Principal Investigator — Assistance Publique - Hôpitaux de Paris (AP-HP), Hôpital Bicètre
Locations (1):
- Hôpital Bicêtre (AP-HP.Université Paris-Saclay), Service de Pneumologie et Soins Intensifs, Le Kremlin-Bicêtre, France, France

IPD SHARING:
Plan to Share IPD: No